CLINICAL TRIAL: NCT06798181
Title: The Effect of Neuropathic Pain on Self-Care Ability and Quality of Life in Type II Diabetic Patients
Brief Title: Neuropathic Pain and Type II Diabetic Patients
Status: Recruiting | Type: Observational
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: Burcu Bayrak 3
Record Dates: First submitted 2024-12-20; First posted 2025-01-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2024-12

CONDITIONS: Neuropathic Pain; Quality of Life; Diabetic Neuropathies
MeSH Terms: conditions — Neuralgia; Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diabetes Mellitus (DM) is a common metabolic disease characterized by hyperglycemia resulting from insufficiency, deficiency or absence of the insulin hormone. Chronic hyperglycemia, secondary metabolic and microvascular changes resulting in diabetic neuropathy are among the most common complications encountered in DM patients.

Diabetic neuropathy is called peripheral, autonomic or spinal depending on the region of involvement. Peripheral involvement is more common than other region involvement and its prevalence in DM patients is observed to be 16-87%. Diabetic peripheral neuropathy (DPN) presents with numbness, tingling, paresthesia, muscle weakness and pain. These symptoms can start from the toes and progress to the leg and even the upper extremities.

In diabetic peripheral neuropathy, pain is seen as burning, electric shock or sharp cold pain, increases at night and affects sleep quality. In these patients, daily living activities such as walking, climbing stairs, and sleeping are negatively affected by progressive DPN and pain, falls are observed, mood disorders are experienced, and the quality of life decreases.

DETAILED DESCRIPTION:
In the study, the Data Descriptive Characteristics Form, Diabetes Quality of Life Scale, Self-Care Efficacy Scale, Neuropathic Symptoms and Signs Self-Assessment Scale and Visual Analog Scale will be used. Data will be collected using face-to-face interview technique with patients who apply to the Internal Medicine Outpatient Clinic and are diagnosed with Type II Diabetes. The researchers will conduct the data collection process between 09:00-16:00 on weekdays. After the patients are informed about the research, their informed consent will be obtained and they will be included in the study.

The Descriptive Characteristics Form was developed by the researchers by reviewing the relevant literature. It consists of 17 questions including information such as age, gender, chronic diseases, and medications used.

The original version of the Diabetes Quality of Life Scale, Diabetes Quality of Life (DQOL) scale was developed in 1988 by the Diabetes Control and Complications Study group.The Turkish culturally compatible version of the DQOL scale consists of four sub-dimensions and a total of 45 questions. The Cronbach α coefficient of the Turkish version of the DQOL scale translated by Yıldırım is 0.89.

Self-Care Agency Scale: The Self-Care Agency Scale was developed in 1979 and was adapted to Turkish in the Republic of Turkey and its validity and reliability were performed. The scale, which focuses on individuals' self-assessment of their involvement in self-care actions, consists of 35 items. The Cronbach Alpha Internal Consistency Coefficient of the scale was found to be 0.89.

VAS-Visual Analog Scale It is a scale divided into equal distances on a 10 cm horizontal plane with no pain on one side and "unbearable" pain on the other side. The patient is asked to mark the point on this line that best expresses the intensity of his/her pain. This distance, measured in millimeters, is interpreted as a "score". For pain intensity, 0 points are evaluated as "no pain" and 10 points as "the worst unbearable pain".

S-LANSS It is used especially in the evaluation of pain types with neuropathic characteristics. - It can be applied easily and quickly at the bedside. It provides the distinction between neuropathic and nociceptive pain. There are 7 items in total, 5 of which are pain questions and 2 of which are allodynia and needle prick test examinations. 0 Its validity and reliability in our country was conducted by Koç in 2008. The Cronbach alpha value of the scale was calculated as 0.74

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older,
* Diagnosed with type II diabetes,
* Reading and writing,
* No physical or psychological communication barriers,
* Can read and speak Turkish,
* Volunteers

Exclusion Criteria:

* Diagnosed with type I diabetes

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals over the age of 18 diagnosed with Type II diabetes
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Neuropathic pain | 15/12/2024-30/07/2025
  Self-Leeds Assessment of Neuropathic Symptoms and Sign (S-LANSS) will be used to assess neuropathic pain types. When the score obtained from this scale consisting of 7 items is >12, neuropathic pain is diagnosed.
the pain severity | 15/12/2024-30/07/2025
  As the first outcome of the study, the patients' neuropathic pain status and pain intensity will be determined. The following scales will be used for this.
  VAS-Visual Analog Scale will be used to assess pain. Scoring will be between 0-10.

SECONDARY OUTCOMES:
Quality of life will be measured with the Diabetes Quality of Life (DQOL) scale | 15/12/2024-30/07/2025
  In the study, the quality of life be measured with the Diabetes Quality of Life (DQOL) scale of life of the patients will be measured with the Diabetes Quality of Life (DQOL) scale. 45 questions will be asked in this scale and the answers will be scored.
the Self-Care Agency Scale | 15/12/2024-30/07/2025
  In addition, the Self-Care Agency of the patients will be evaluated. For this, the Self-Care Agency Scale will be used. This scale consists of 35 items. As the score obtained from the scale increases, the self-care agency increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Seyh Edeabli University, Bilecik, Turkey (Türkiye)